CLINICAL TRIAL: NCT05427968
Title: To Tilt or Not to Tilt?: Comparison of Severity of Hypotension Between Supine and Left Tilt Position During Spinal Anesthesia for Elective C-section
Brief Title: Comparison of Hypotension During Spinal Anaesthesia for C-section
Status: Completed | Type: Observational
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Rubaid Azhar Dhillon, MBBS, Rawalpindi Medical College
Other Study IDs: 2021-4711-17843
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Hypotension; Cesarean Section; Aortocaval Compression
Keywords: Hypotension; Cesarean Section; Aortocaval Compression; Left titl
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supine group: Spinal anaesthesia was administered in sitting position and then supine position was maintained.
- Left tilt group: Spinal anesthesia was administered in sitting position was then maintained on supine position until full anesthetic effect (motor and sensory loss) and then table was tilted 15 degrees to the left.

SUMMARY:
Maternal hypotension during C section has been reported due to aortocaval compression (ACC) by full term uterus in supine position. This study aimed at reporting the effect of left tilt on maternal hemodynamics.

DETAILED DESCRIPTION:
C-section is usually done in either general anesthesia or regional (epidural or spinal) anesthesia. The choice lies with the mother. In spinal anesthesia the anaesthetic agent is injected into the subarachnoid space. Hypotension in supine position that is associated with full term gravid uterus has been explained by compression of inferior venacava (IVF) and aorta. This aortocaval compression (ACC) can also cause hypotension during C- section after spinal block.

The aim of our study was to study the effect of left tilt on systolic (SBP) and diastolic blood pressure (DBP), heart rate and the frequency of phenylephrine used to maintain the blood pressure in normal range.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years, undergoing Elective Caesarean Section for term singleton pregnancy, ASA I/II, were included after their consent for the participation of the study.

Exclusion Criteria:

* Participants with co-morbidities (Hypertension, diabetes mellitus, cardiovascular or cerebrovascular disease and a history of coagulation disorders), any contraindication to spinal anesthesia, with multiple pregnancy, pre-eclampsia, obesity (body mass index > 30 kg.m2), intrauterine growth were excluded from the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only females included undergoing C-section
Study Population: Participants after fulfilling the inclusion exclusion criteria were randomized by lottery method into two groups; supine group (Group 1) and left tilt group. (Group 2).
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Group 1 - Supine Group | December 2021 to February 2022
  Systolic blood pressures decreased significantly in the supine group
Group 2 - Left tilt Group | December 2021 to February 2022
  The decrease in the diastolic blood pressure was marginally significant in the left tilt group.

CONTACTS AND LOCATIONS:
Locations (1):
- Rawalpindi Medical University, Rawalpindi, Punjab Province, Pakistan